CLINICAL TRIAL: NCT01204788
Title: A Prospective Randomized Comparative Study of the Effect on Infections of Radiated Prophylactic White Cell Transfusions Versus Therapeutic Radiated White Cell Transfusions
Brief Title: Prophylactic White Cell Transfusions Versus Therapeutic White Cell Transfusions in Patients With Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Recruitment
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010-0468; NCI-2012-01795 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-05

CONDITIONS: Leukemia
Keywords: Acute myelogenous leukemia; AML; Undifferentiated and bi-phenotypic leukemia; High-risk myelodysplastic syndrome; Chronic myelogenous leukemia; Infection; Radiated Prophylactic White Cell Transfusions; Therapeutic Radiated White Cell Transfusion; prophylactic antibiotics
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Disorders of Sex Development; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Prophylactic Arm) (Experimental): Prophylactic Treatment (standard of care prophylactic antibiotics) + Prophylactic White Cell Transfusion
  Interventions: Procedure: Prophylactic White Cell Transfusion
- Arm 2 (Therapeutic Arm) (Experimental): Prophylactic Treatment (standard of care prophylactic antibiotics) + Therapeutic White Cell Transfusion
  Interventions: Procedure: Therapeutic White Cell Transfusion

INTERVENTIONS:
Procedure: Prophylactic White Cell Transfusion — Radiated white blood cell transfusions 2-3 times each week, or daily if infection develops
  Arms: Arm 1 (Prophylactic Arm)
Procedure: Therapeutic White Cell Transfusion — Radiated white blood cell transfusions daily only with infection (or persistent fever)
  Arms: Arm 2 (Therapeutic Arm)

SUMMARY:
Patients with leukemia often have low white blood cell counts after chemotherapy, which puts them at greater risk for infection. The standard of care for preventing infections is to give these patients antibiotic, antifungal, and antiviral drugs during the time that white blood cell counts are low. However, many patients still develop infections during chemotherapy. Radiated white blood cell transfusions are a standard treatment once a patient develops a severe infection.

The goal of this clinical research study is to learn if giving unirradiated white blood cell transfusions early in chemotherapy might delay or prevent infections in patients with leukemia. Researchers also want to learn more about the type and severity of any infections that do occur.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part of this study, and you are 1 of the first 60 participants to be enrolled, you will be randomly assigned (as in the flip of a coin) to 1 of 2 groups:

* If you are in Group 1, you will receive the standard of care drugs that are used to prevent infections. You will also receive unirradiated white blood cell transfusions 2-3 times each week. If at any point you develop an infection, white blood cell transfusions will then be given daily in addition to the standard treatment for the infection.
* If you are in Group 2, you will receive the standard of care drugs that are used to prevent infections. You will only receive unirradiated white blood cell transfusions if at any point you develop an infection. You will receive these transfusions daily, in addition to the standard treatment for the infection.

If you are not 1 of the first 60 participants to be enrolled, you will be assigned to the study group that the study doctor decides is in your best interest. This will be decided based on how the first participants have responded to the different treatments.

The drugs you receive as part of the standard therapy will be up the study doctor.

Study Procedures:

During each white blood cell transfusion, you will receive white blood cells from a volunteer donor through a needle in your vein. Each transfusion will take anywhere from 1 hour to several hours, depending on how you tolerate the treatment.

Before each white blood cell transfusion, your vital signs will be recorded. During and for 1 hour after the transfusion, you will be monitored for side effects. You may be given a drug to help or reduce any side effects. Your doctor will tell you more about any drug that is given for side effects.

While you are in the hospital for leukemia treatment, blood (about 1 teaspoon) will be drawn to check for fungal infections 2-3 times each week. This test will be done 1 time each week when you are not in the hospital until the doctor no longer thinks it is needed.

If at any point you develop a fever while on study, blood (about 1 teaspoon) will be drawn to check for infection. You will also have a CT scan within 3 days of developing a fever. If the doctor thinks it is needed, you will then have a CT scan 2 weeks later and at any other point that the doctor thinks it is needed to check for infection.

Length of Study:

You will continue to have transfusions until the doctor thinks infection has been controlled or until your white blood cell counts stay at a certain level for at least 2 days in a row. If at any point you are discharged from the hospital and your doctor wants you to continue receiving white blood cell transfusions, you will be able to receive them as an outpatient.

You will be monitored for side effects and signs of infection for up to 2 cycles of anti-leukemia treatment through a review of your medical record. You will be taken off study if you have intolerable side effects.

This is an investigational study. Radiated white blood cell transfusions are considered to be a standard procedure for the treatment of serious infections. It is investigational to give unirradiated white blood cell transfusions as a way of preventing infections.

Up to 240 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Adult and pediatric (=/> 2 years old) patients with a diagnosis of acute myelogenous leukemia (including undifferentiated and bi-phenotypic leukemia), or high-risk myelodysplastic syndrome, or chronic myelogenous leukemia in blast crisis who will receive first or second anti-leukemia therapeutic intent with chemotherapy, targeted therapy or hypomethylating agents
2. Patients must sign an informed consent indicating they are aware of the investigational nature of this study, in keeping with the policies of the hospital.

Exclusion Criteria:

1. Patients with baseline (at start leukemia treatment) infection, defined as patients with a)fever and known positive cultures at the time of randomization; or b) chest or sinus computed tomography with findings suggestive of pneumonia or sinusitis; or c) one positive galactomannan test >/= 1 or two positive galactomannan text >/= 0.5 to 1
2. Patients with Zubrod performance status >/= 3

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emil J Freireich, MD, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 15, 2010 to January 2, 2013. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: One participant was not treated and is therefore excluded from the trial.
Groups:
- Arm 1 (Prophylactic Arm): Prophylactic Treatment (standard of care prophylactic antibiotics) + Prophylactic White Cell Transfusion. Radiated white blood cell transfusions 2-3 times each week, or daily if infection develops
- Arm 2 (Therapeutic Arm): Prophylactic Treatment (standard of care prophylactic antibiotics) + Therapeutic White Cell Transfusion. Radiated white blood cell transfusions daily only with infection (or persistent fever)
Period: Overall Study
Arm/Group | Arm 1 (Prophylactic Arm) | Arm 2 (Therapeutic Arm)
Started | 1 | 3
Completed | 0 | 0
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Prophylactic Arm) | Arm 2 (Therapeutic Arm) | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Infection
Description: Primary outcome is infection (yes/no) where participant without infection found by day 42 patient are counted as 'No' to infection.
Time Frame: Blood draw 2-3 times a week while hospitalized, weekly thereafter. Participant to remain on study 42 days after transfusion.
Population: Outcomes inevaluable due to low recruitment.
Arm/Group | Arm 1 (Prophylactic Arm) | Arm 2 (Therapeutic Arm)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected for up to two cycles of anti-leukemia treatment. Overall study period: June 16, 2011 to August 30, 2012.
Arm/Group | Arm 1 (Prophylactic Arm) | Arm 2 (Therapeutic Arm)
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes